CLINICAL TRIAL: NCT04460521
Title: The Use of N-acetylcysteine Supplementation in Addition to Night Splinting for Treatment of Mild to Moderate Carpal Tunnel Syndrome: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: The ACTS Trial: N-acetylcysteine (NAC) and Night-splinting as a Non-operative Treatment for Carpal Tunnel Syndrome
Acronym: ACTS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emily Krauss (Other)
Responsible Party: Sponsor-Investigator, Emily Krauss, Physician, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTS Trial
Record Dates: First submitted 2020-06-17; First posted 2020-07-07 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Carpal Tunnel Syndrome; Hand Injuries and Disorders; Nerve Compression; Splints; Carpal Tunnel; Carpal Tunnel Release
Keywords: Wrist splint; Carpal tunnel syndrome; Carpal tunnel release; Compression neuropathy; NAC; Conservative treatment; Hand surgery; Plastic surgery; N-acetylcysteine; Night splint
MeSH Terms: conditions — Carpal Tunnel Syndrome; Hand Injuries; Disease; Neuroma; Median Neuropathy; Tomaculous neuropathy | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will undergo permutated block randomization to either the placebo controlled or experimental group in a 1:1 ratio. This method will be computer-generated. The allocation sequence will be concealed to research staff. The participants, clinic nurses, research assistants, and physician investigators as well as outcome assessors will be masked to participant group allocation. Unblinding will be permissible in extenuating circumstances only, such as if a participant experiences a severe adverse reaction secondary to the tablet and requires confirmation of the contents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NAC Group (Experimental): Participants in this group will given an N-acetylcysteine 500mg oral tablet daily in addition to wearing a standard carpal tunnel splint nightly (worn approximately 6-8 hours/day). Both interventions will take place concurrently for a total of 8 consecutive weeks.
  Interventions: Drug: N-Acetyl cysteine; Device: Wrist Splint
- Placebo Group (Placebo Comparator): Participants in this group will be given a placebo table to be taken orally daily in addition to wearing a standard carpal tunnel splint nightly (worn approximately 6-8 hours/day). Both interventions will take place concurrently for a total of 8 consecutive weeks.
  Interventions: Device: Wrist Splint

INTERVENTIONS:
Drug: N-Acetyl cysteine — In addition to splinting, both groups will receive an oral tablet to take daily for 8 weeks. Participants assigned to the experimental group will receive oral NAC (500 mg PO daily for eight weeks; based on recommended daily dose for use as an antioxidant and dosing in previous human clinical trials and animal studies), and those assigned to the control group will be given a similar looking placebo with identical instructions. Tablets will be provided in a blister pack to assist with compliance.
  Arms: NAC Group
Device: Wrist Splint — Participants in both arms will be given a standard prescription for a prefabricated night splint which keeps the wrist in a neutral position and instructed on proper use and the importance of consistent use. To limit splint variability, we will ensure that splint prescriptions are written such that a MedSpec Wrist Lacer II splint is obtained from the patient's pharmacy. This is the most commonly available brand locally and meets the criteria for wrist, metacarpophalangeal, and interphalangeal joint positioning. They will be advised to wear the splint consistently during sleeping hours on their affected wrist for eight weeks, as is the standard of practice.

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common nerve compression syndrome worldwide, causing significant chronic pain, functional impairment, and lowered quality of life for individuals of various backgrounds. CTS is caused by chronic compression of the median nerve in the carpal tunnel of the wrist, causing numbness and pain in the palm, thumb, index, and middle fingers and eventual weakness of the hand. Many different treatments for CTS have been proposed and studied, including but not limited to non-operative treatments such as wrist splinting, steroid injections, and lifestyle modifications as well as operative treatments, such as surgical carpal tunnel release (CTR). To date, very few oral medications have been shown to be effective as conservative treatments for CTS. In this study the investigators will examine whether there is any benefit to using oral N-acetylcysteine (NAC) as an adjunctive treatment for mild to moderate CTS in addition to a standard 8-week trial of night splinting. NAC has been used in humans for various purposes, is extremely safe and has very few side effects, and has been shown to have anti-inflammation properties which may help treat CTS. The investigators will study this by performing a randomized controlled trial, comparing patients receiving oral NAC and standard night splinting to patients receiving an identical placebo and standard night splinting. Both patient groups will be assessed using a questionnaire to assess for severity of their CTS symptoms both before and after the 8-week treatment. The primary objective will be to determine whether supplementation with oral NAC in addition to night splinting has any significant impact on patient-reported symptoms and functional impairment when compared to night splinting alone. The investigators will also measure secondary outcomes including whether patients decide to have surgery for their CTS after treatment and/or continued use of other treatments. This study has the potential to have a significant positive impact on patients by identifying a safe, inexpensive, accessible, and well tolerated conservative treatment for mild to moderate carpal tunnel syndrome, and potentially preventing the need for additional, more invasive treatments such as surgery.

DETAILED DESCRIPTION:
Introduction: Carpal tunnel syndrome (CTS) is the most prevalent and widely studied peripheral nerve entrapment syndrome, with estimates between 10-20% of the general population having clinical symptoms of CTS at least once in their lifetime. Classically, it presents with symptoms of nocturnal numbness and tingling in the distribution of the median nerve, often progressing to more constant parasthesias, weakness, and pain in the hand and/or wrist, and eventually thenar muscle atrophy. There is a robust and continuously growing body of research available on the clinical presentation, diagnosis, and management of CTS. Conservative, non-operative management strategies, including night splinting and corticosteroid injections, have shown significant clinical benefit in improving the severity of CTS symptoms and preventing the need for carpal tunnel release (CTR) surgery. However, many patients with mild-moderate CTS will still go on to have CTR due to failure of conservative measures or lack of long-term efficacy. N-acetylcysteine (NAC) is a safe and extremely well tolerated compound which acts as a powerful antioxidant and has been utilized in the treatment of many conditions including, but not limited to acetaminophen toxicity, various psychiatric disorders, Alzheimer's disease, and polycystic ovarian syndrome. Of note, some studies using animal models have shown NAC to be effective in reducing oxidative stress and potentially expediting the recovery of peripheral nerve injuries. This warrants consideration of the potential of NAC to impact peripheral nerve recovery in the non-operative treatment of mild to moderate carpal tunnel syndrome. Given the safety of NAC, and promising hypotheses to suggest neuroprotective and neuronal growth promoting effects on peripheral nerves, The investigators propose the following project to examine whether supplementation with oral NAC in addition to standard night splinting significantly improves functional outcomes for mild to moderate CTS when compared to splinting alone.

Methods: This study will be a randomized, double-blind, parallel-group, placebo-controlled human clinical trial. Participants for this study will be recruited by staff, residents, and research assistants on a voluntary basis from both the outpatient Plastic Surgery clinic, Plastic Surgery clinic waiting list, and the Neurology clinic at the Queen Elizabeth II Health Sciences Center, Halifax Infirmary, in Nova Scotia, Canada. These will include patients both waiting for consultation with a hand surgeon for consideration of carpal tunnel release and patients who have already been assessed by a hand surgeon but have yet to undergo a trial of night splinting.

For the purposes of this study, a diagnosis of mild to moderate CTS will be primarily determined by clinical history of any intermittent or persistent numbness in the distribution of the median nerve and/or pain in the hand or wrist. Clinical exam findings consistent with a diagnosis of CTS will be determined by a CTS-6 score of 12 or higher, indicating at least an 80% chance of a diagnosis of CTS.

After identification of eligible participants, they will be informed of the nature of the study and the proposed intervention and consented both verbally and in writing to participate in the study by a research assistant. They will undergo permutated block randomization to either the placebo controlled or experimental group in a 1:1 ratio. The participants and physicians/assessors will be masked to participant group allocation.

Baseline variables will be collected from each participant including age, gender, smoking status, previous diagnoses of carpal tunnel syndrome, which side is affected or bilateral disease, which side will undergo splinting as determined by severity, previous treatments for carpal tunnel syndrome on both the study and non-study limb (if bilateral disease), clinical and electrodiagnostic severity of CTS, duration of symptoms, nature of onset, any current pain medications for both CTS symptoms and non-CTS related pain, employment status, and comorbidities.

Pre-treatment Evaluation: Once the participants have given informed consent and been randomized, they will be asked to complete a baseline Boston Carpal Tunnel Questionnaire (BCTQ). All patients will receive a prescription for a wrist splint and 8 weeks supply of either NAC tablets or a placebo.

Post-treatment Evaluation: Follow-up will take place at eight weeks by the surgeon to whom the patient was referred for consideration of carpal tunnel release. Participants will be asked to complete another BCTQ to be compared to their baseline score. At this time, patients can decide if they wish to proceed with carpal tunnel release surgery or defer surgical treatment.

For patients that do not decide to proceed with carpal tunnel release surgery, a secondary outcome measure will include a follow up at 6 months, at which time The investigators will collect patient reported outcomes including conversion to surgery, continued use of conservative treatment modalities including night splinting or other treatment modalities, and patient-reported outcomes in the way of a final BCTQ if surgery was not pursued.

Outcome Measures: The primary outcome measure in this study will be the overall score for symptom severity and hand function limitations as determined by the BCTQ at eight weeks post initiation of night splinting therapy. A secondary outcome will be ratio of conversion to surgery versus continuation of conservative treatment or no treatment at all.

Data Analysis: For baseline demographic variables, The investigators will use descriptive statistics (means with standard deviations for continuous variables or frequency with percentages for categorical variables) and assess between group similarities. T-test and chi-square tests, where appropriate, will be used to determine significant differences in baseline demographics. The primary between group analysis will be done with multiple linear regression with adjustments made for age at randomization, gender, symptom duration, and baseline BCTQ score, with an aim to identify significant differences in improvements in the BCTQ score between the treatment and control group at eight weeks and six months, where applicable. The investigators will also examine for significance in the ratio of conversion to surgery at eight weeks and six months. Significance will be set as a p-value <0.05.

Sample Size: Based on the INSTINCTS trial by Chesterson and colleagues, this study will require 240 total participants (120 per group). The investigators will aim to detect a 15% or greater improvement in the BCTQ from assumed baseline value of 2.9 (scale 1-5, SD 1.0). This would mean a 0.9 point (30%) reduction in the NAC plus splinting group and a 0.45 point (15%) reduction in the placebo plus splinting group, with a pooled SD of 1.0 and mean difference of 0.45. Power will be set at 90%, two-tailed significance at 5%, and a 15% loss to follow up will be anticipated. Recruitment of 120 participants for both the placebo-controlled and NAC groups will primarily be from the practice of a single hand surgeon (DT) and the practices of several local neurologists. The primary hand surgeon (DT) has completed a preliminary audit of his practice and has determined that in the last year, he completed 200 CTRs in the minor procedure clinic.

Strengths and Limitations: This study will have a robust sample size, minimal potential for participant loss, and strong clinical applications in the way of a minimally invasive adjunct to night splinting as a conservative treatment for mild to moderate carpal tunnel syndrome. This study is limited in that the primary outcome measure is relatively subjective, despite the fact that the BCTQ is a validated tool that has been applied clinically in reputable trials. Additionally, despite controlling for between group variability in baseline function, severity of disease prior to treatment can certainly impact the degree of response to conservative measures and may confound results.

Ethical Considerations: Given that the participants in this study will have already decided to pursue investigations and treatment for their carpal tunnel syndrome prior to being informed of and consented for our trial, there is a negligible ethical conflict of exposing a patient to tests and treatments that they would not have otherwise had. Eligible participants will be given the standard information regarding the risks and benefits of both pursuing and delaying carpal tunnel release surgery and will not be delayed or denied surgery should they choose not to participate in the trial. It is, however, acknowledged that there is a remote possibility of placing patients at risk by administering a medication. NAC has been found to be a safe, non-toxic substance with little-to-no reported short or long-term side effects. Participants will be given as much information about the possible intervention as is needed and will be offered the right to withdraw from the study at any point in time without any repercussion to their medical care.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a confirmed diagnosis of mild to moderate idiopathic unilateral or bilateral CTS as determined by both clinical exam findings and electrodiagnostic nerve conduction studies (median nerve distal motor latency ≥ 4.3 milliseconds and/or median nerve sensory distal latency ≥ 3.5 milliseconds at the wrist) performed within the preceding year prior to enrollment
2. Symptoms of CTS must have been present for ≥ 6 weeks
3. The patient must be ≥ 18 years of age.

Exclusion Criteria:

1. Any previous carpal tunnel release procedure on the ipsilateral limb
2. Any previous corticosteroid injection in the last 6 months on the ipsilateral limb
3. Severe CTS/signs of median nerve denervation with axonal loss determined by constant wrist or hand pain, constant parasthesias in the median nerve distribution, or thenar muscle atrophy in the ipsilateral limb
4. Any known or suspected allergy to NAC
5. Any current medications which preclude use of NAC including antibiotics or nitroglycerin
6. Breastfeeding patients or patients with nephrolithiasis
7. Any history of proximal ipsilateral neck or proximal limb injury
8. Secondary CTS related to pregnancy
9. Unable for financial reasons to obtain a night splint (i.e. lack of insurance coverage or lack of financial means).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Boston Carpal Tunnel Questionnaire (BCTQ) at 8 weeks | 8 weeks
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a validated tool for patient-reported outcomes with respect to symptoms and functional impact of carpal tunnel syndrome. It consists of both a symptom severity scale (SSS) (11 items) and functional status scale (FSS) (8 items). Each item on both of these scales is scored on a 5-point rating system, with higher numbers indicating more severe symptoms and higher functional disability. The possible range of both the FSS and SSS combined is from 19-95. A baseline BCTQ will be administered at the first visit, which will be used to calculate the overall change in BCTQ score at 8 weeks.

SECONDARY OUTCOMES:
Number of participants who elect to have surgical carpal tunnel decompression after 8 weeks | 8 weeks
  The participant's decision to continue with conservative treatment or to elect to have a carpal tunnel release procedure at 8-weeks post-treatment will be a secondary outcome measure.
Number of participants who elect to have surgical carpal tunnel decompression after 6 months | 6 months
  If at 8-weeks, the participant decides not to have carpal tunnel release surgery, an additional follow up visit will be scheduled at 6 months time. At this point in time, the participants decision to have carpal tunnel release surgery or to continue to conservative modalities will be a subgroup analysis.
Change from baseline Boston Carpal Tunnel Questionnaire (BCTQ) at 6 months | 6 months
  If the participant decides not have have a carpal tunnel release at 8 weeks, an additional follow up visit will be scheduled in 6 months. At this time, a third BCTQ will be completed to assess change in long-term BCTQ compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD, Study Director — NSHA
Locations (1):
- Queen Elizabeth II Health Sciences Center, Halifax Infirmary Site, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Background] Chesterton LS, Blagojevic-Bucknall M, Burton C, Dziedzic KS, Davenport G, Jowett SM, Myers HL, Oppong R, Rathod-Mistry T, van der Windt DA, Hay EM, Roddy E. The clinical and cost-effectiveness of corticosteroid injection versus night splints for carpal tunnel syndrome (INSTINCTS trial): an open-label, parallel group, randomised controlled trial. Lancet. 2018 Oct 20;392(10156):1423-1433. doi: 10.1016/S0140-6736(18)31572-1. PMID 30343858
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Mokhtari V, Afsharian P, Shahhoseini M, Kalantar SM, Moini A. A Review on Various Uses of N-Acetyl Cysteine. Cell J. 2017 Apr-Jun;19(1):11-17. doi: 10.22074/cellj.2016.4872. Epub 2016 Dec 21. PMID 28367412
- [Background] Huisstede BM, Friden J, Coert JH, Hoogvliet P; European HANDGUIDE Group. Carpal tunnel syndrome: hand surgeons, hand therapists, and physical medicine and rehabilitation physicians agree on a multidisciplinary treatment guideline-results from the European HANDGUIDE Study. Arch Phys Med Rehabil. 2014 Dec;95(12):2253-63. doi: 10.1016/j.apmr.2014.06.022. Epub 2014 Aug 12. PMID 25127999
- [Background] Page MJ, Massy-Westropp N, O'Connor D, Pitt V. Splinting for carpal tunnel syndrome. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD010003. doi: 10.1002/14651858.CD010003. PMID 22786532
- [Background] Chan KM, Gordon T, Zochodne DW, Power HA. Improving peripheral nerve regeneration: from molecular mechanisms to potential therapeutic targets. Exp Neurol. 2014 Nov;261:826-35. doi: 10.1016/j.expneurol.2014.09.006. Epub 2014 Sep 16. PMID 25220611
- [Background] Reid AJ, Shawcross SG, Hamilton AE, Wiberg M, Terenghi G. N-acetylcysteine alters apoptotic gene expression in axotomised primary sensory afferent subpopulations. Neurosci Res. 2009 Oct;65(2):148-55. doi: 10.1016/j.neures.2009.06.008. Epub 2009 Jun 24. PMID 19559059
- [Background] Sud V, Freeland AE. Biochemistry of carpal tunnel syndrome. Microsurgery. 2005;25(1):44-6. doi: 10.1002/micr.20071. PMID 15481038
- [Background] Kim JK, Koh YD, Kim JS, Hann HJ, Kim MJ. Oxidative stress in subsynovial connective tissue of idiopathic carpal tunnel syndrome. J Orthop Res. 2010 Nov;28(11):1463-8. doi: 10.1002/jor.21163. PMID 20872582
- [Background] Lingjaerde O, Ahlfors UG, Bech P, Dencker SJ, Elgen K. The UKU side effect rating scale. A new comprehensive rating scale for psychotropic drugs and a cross-sectional study of side effects in neuroleptic-treated patients. Acta Psychiatr Scand Suppl. 1987;334:1-100. doi: 10.1111/j.1600-0447.1987.tb10566.x. No abstract available. PMID 2887090